CLINICAL TRIAL: NCT06987851
Title: An Extension, Multicenter, Open-Label, Non-Comparative Clinical Study of the Efficacy and Safety of Long-Term Use of BCD-132 (JSC BIOCAD) in Patients With Multiple Sclerosis Who Previously Received Therapy in Clinical Studies of JSC BIOCAD
Brief Title: An Extension Clinical Study of the Efficacy and Safety of BCD-132 in Patients With Multiple Sclerosis Who Previously Received Therapy in Clinical Studies of JSC BIOCAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-132-EXT
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis, relapsing multiple sclerosis, anti-CD20, DMT, divosilimab
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCD-132 (divozilimab) (Experimental): Intravenous infusion of BCD-132 every 24 weeks
  Interventions: Biological: Divozilimab

INTERVENTIONS:
Biological: Divozilimab — Intravenous infusion of BCD-132 every 24 weeks

SUMMARY:
The aim of this clinical study is to assess the long-term efficacy and safety of BCD-132 (divozilimab) in patients with multiple sclerosis who previously participaded in BCD-132-2 and BCD-132-4/MIRANTIBUS studies

DETAILED DESCRIPTION:
Clinical study BCD-132-EXT is a Phase III study extension conducted after completion of BCD-132 500 mg therapy by subjects of clinical studies BCD-132-2 and BCD-132-4/MIRANTIBUS.

The study is designed as a multicenter, open-label, non-randomized, non-comparative, single-arm clinical study.

The study consists of a screening period (14 days), a treatment period (96 weeks) and a follow-up period (4 weeks). During treatment period, the subjects will receive the investigational product BCD-132 (divozilimab).

The duration of participation for each subject will be approximately 102 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the subject to participate in the study has been obtained.
* The subject was in the BCD-132 500 mg group in BCD-132-2, then transferred to BCD-132-4/MIRANTIBUS and completed it according to the Protocol (completed all scheduled study visits).
* Last administration of BCD-132 in BCD-132-4/MIRANTIBUS was performed at least 22 weeks before the planned date of the first drug administration in this clinical study.

Exclusion Criteria:

* Heart failure (NYHA class III/IV).
* Malignancies detected after completion of study BCD-132-4/MIRANTIBUS and prior to signing the informed consent to participate in this study, as well as conditions (acute and chronic) precluding further treatment and participation in the study in the Investigator's opinion.
* Metabolic abnormalities according to blood chemistry (including increased creatinine, urea, ALT, AST) and/or blood count abnormalities (including decreased white blood cell count, absolute lymphocyte count, absolute neutrophil count, platelet count, decreased hemoglobin concentration) identified at the screening and precluding further treatment and participation in the study in the Investigator's opinion.
* Pregnancy, breastfeeding, or planned pregnancy at any time during the participation in the study and 48 weeks after the scheduled last administration of the product in this study.
* Use, between the completion of participation in BCD-132-4/MIRANTIBUS and the signing of the informed consent for this study, of the following drugs: anti-B cell therapies (e.g., rituximab, ocrelizumab, abatacept, belimumab, ofatumumab, and others); alemtuzumab, daclizumab, teriflunomide, mitoxantrone, cladribine; cyclophosphamide, cyclosporine, azathioprine; mycophenolate mofetil, fingolimod and other sphingosine-1-phosphate (S1P) receptor modulators, natalizumab.
* Known intolerance, including hypersensitivity to any component of BCD-132, premedication drugs, or conditions in which the above drugs are contraindicated in the Investigator's opinion.
* Historical evidence of progressive multifocal leukoencephalopathy (PML).
* Contraindications to MRI and the use of gadolinium-containing contrast agents, including, but not limited to, the presence of metal foreign bodies, artificial heart valves, electronic middle ear implants, pacemakers; allergies to gadolinium or gadolinium-containing contrast agents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Annualized relapse rate | 48 and 96 weeks

SECONDARY OUTCOMES:
Time to first relapse | 102 weeks
Proportion of patients without confirmed relapses | 48 and 96 weeks
Total number of T1 Gd+ lesions (per scan) | 48 and 100 weeks
Proportion of patients without contrast-enhancing lesions | 48 and 100 weeks
Proportion of patients without new or enlarging T2 lesions | 48 and 100 weeks
Number of new or enlarged T2 lesions | 48 and 100 weeks
Number of CUA (Combined Unique Active) lesions | 48 and 100 weeks
  Total number of new contrast-enhancing T1 lesions and new T2 lesions or enlarged T2-weighted lesions without double counting on MRI (Combined Unique Active)
Changes over time in neurological deficit parameters according to the Expanded Disability Status Scale (EDSS) | 102 weeks
Changes over time in Timed 25-Foot Walk Test | 102 weeks
Changes over time in 9-Hole Peg Test | 102 weeks
Changes over time in Symbol Digit Modalities Test (SDMT) | 102 weeks
Changes over time in quality of life indicators assessed with the SF-36 questionnaire | 102 weeks

CONTACTS AND LOCATIONS:
Locations (15):
- Russia (15):
  - Vyacheslav Andreyevich Dudin, Kirov
  - Dmitry Vladimirovich Pokhabov, Krasnoyarsk
  - Ivan Aleksandrovich Shchukin, Moscow
  - Sergey Viktorovich Kotov, Moscow
  - Elena Vladimirovna Parshina, Nizhny Novgorod
  - Irina Aleksandrovna Sokolova, Nizhny Novgorod
  - Gennady Nikolayevich Mishin, Pyatigorsk
  - Yuri Vladimirovich Trinitatsky, Rostov-on-Don
  - Zoya Aleksandrovna Goncharova, Rostov-on-Don
  - Leonid Grigoryevich Zaslavsky, Saint Petersburg
  - Natalya Agafonovna Totolyan, Saint Petersburg
  - Irina Yevgenyevna Poverennova, Samara
  - Valentina Mikhaylovna Alifirova, Tomsk
  - Stella Anatolyevna Sivertseva, Tyumen
  - Irina Vladimirovna Greshnova, Ulyanovsk

IPD SHARING:
Plan to Share IPD: No